CLINICAL TRIAL: NCT03638973
Title: Randomized Prospective Study for the Comparison of Sample Biopsy Using Scalpel or Er:YAG Laser
Brief Title: Comparison of Sample Biopsy Using Scalpel or Er:YAG Laser
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018-01364
Record Dates: First submitted 2018-08-13; First posted 2018-08-20 (Actual); Last update posted 2018-10-12 (Actual); Status verified 2018-10

CONDITIONS: Laser Burn; Gingival Disease; Biopsy Wound
MeSH Terms: conditions — Gingival Diseases | interventions — Biopsy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Biopsy with Er: YAG (Experimental): Removal of specimen biopsies in patients with leukoplakic or lichenoid mucosal lesions using Er: YAG laser under previous local anesthesia
  Interventions: Procedure: Biopsy
- Biopsy with Scalpel (Active Comparator): Biopsies taken with Er: YAG are compared with biopsies taken with a scalpel in patients with lichenoid or leukoplakic changes of the oral mucosa.
  Interventions: Procedure: Biopsy

INTERVENTIONS:
Procedure: Biopsy — Removal of specimen biopsies in patients with leukoplakic or lichenoid mucosal lesions using Er: YAG laser or scalpel under previous local anesthesia.

SUMMARY:
For certain changes in the oral mucosa a histopathological examination of the affected tissue is indicated to confirm the diagnosis. The gold standard is the biopsy by scalpel. The aim of this study is to compare the alternative method of tissue sampling using the erbium doped yttrium aluminium garnet (Er:YAG) laser with the gold Standard.

DETAILED DESCRIPTION:
Various parameters are compared, such as the pain intensity during and after the biopsy, the evaluation of the tissue removed by the histopathologist, the occurrence of bleeding during and after the removal and the time required for both therapies.

Patients who agree to participate in the study will be randomized (randomly) to either therapy.

ELIGIBILITY:
Inclusion Criteria:

* Indication for biopsy of the oral mucosa
* male and female adult patients
* Written consent of the participating persons after clarification

Exclusion Criteria:

* pregnancy
* Taking blood thinners
* Known infectious diseases
* Untreated diabetes mellitus
* Taking immunosuppressants

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2018-11-01 (Estimated); Primary Completion 2019-11-01 (Estimated); Study Completion 2020-11-01 (Estimated)

PRIMARY OUTCOMES:
histological assessability | 13 month
  The primary endpoint is the histological assessability of the samples. This is evaluated by the histologist and divided into degrees 0-3. The
  Subdivision of the artifacts takes place according to the following degrees:
  0: none, 1: slight artifacts, not affecting the evaluation of the sample, 2: moderate artifacts, slight deterioration in the evaluability of the sample, 3: severe artifacts, severely impaired

SECONDARY OUTCOMES:
postoperative pain | 13 month
  The pain is measured by the visual analogue scale (VAS) 0-10, 0 = no pain, 10 = worst possible pain
postoperative bleeding | 13 month
  The bleeding is determined with yes or no.
time for removal | 13 month
  The time to remove is measured in seconds

CONTACTS AND LOCATIONS:
Overall Officials: Martin Rücker, Prof.Dr.Dr., Principal Investigator — Sponsor GmbH
Locations (1):
- Clinic for Oral Surgery, Center of dental medicine, University of Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Suter VGA, Altermatt HJ, Bornstein MM. A randomized controlled clinical and histopathological trial comparing excisional biopsies of oral fibrous hyperplasias using CO2 and Er:YAG laser. Lasers Med Sci. 2017 Apr;32(3):573-581. doi: 10.1007/s10103-017-2151-8. Epub 2017 Jan 24. PMID 28120248